CLINICAL TRIAL: NCT01142011
Title: A Single Arm, Phase II Study of the Anti-Blys Monoclonal Antibody, Belimumab in Symptomatic Waldenstroms Macroglobulinaemia
Brief Title: A Study of Belimumab in Treating Symptomatic Waldenstroms Macroglobulinaemia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cancer Trials Australia (Other)
Collaborators: Human Genome Sciences Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HGSI Belimumab in WM
Record Dates: First submitted 2010-06-10; First posted 2010-06-11 (Estimated); Last update posted 2012-02-10 (Estimated); Status verified 2012-02

CONDITIONS: Symptomatic Waldenstroms Macroglobulinaemia
Keywords: Waldenstroms; Belimumab; anti Blys; monoclonal antibody
MeSH Terms: interventions — belimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Belimumab (Experimental): The first cycle of Belimumab is a loading cycle of 3 doses over 28 days (days 1, 15, 29).
  After the first cycle, additional cycles of belimumab will be administered every 28 ± 1 days (cycle 2 and all subsequent cycles).
  Interventions: Drug: Belimumab

INTERVENTIONS:
Drug: Belimumab — The first cycle of Belimumab (10mg/kg by intravenous (IV) infusion) is a loading cycle of 3 doses over 28 days (days 1, 15, 29). After the first cycle, additional cycles of belimumab (10mg/kg by intravenous (IV) infusion) will be administered every 28 ± 1 days (cycle 2 and all subsequent cycles).
  The infusion will be administered over a minimum period of 1 hour.

SUMMARY:
Hypothesis; That inhibition of plasma Blys by the monoclonal antibody Belimumab will reduce both the survival of the lymphoplasmacytoid cells of Waldenstrom Macroglobulinaemia (WM), and their production of monoclonal IgM, resulting in a reduction of IgM paraprotein.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age.
* Diagnosis of WM histologically confirmed on bone marrow biopsy.
* Detectable IgM paraprotein >5 g/L
* Less than 3 lines of prior therapy for WM
* Full blood count within 4 weeks prior to screening shows ANC >1.0 x109/l AND platelet count >50 x109/l
* Therapy indicated due to development of one or more of the following:

  1. symptomatic anaemia
  2. hyperviscosity symptoms
  3. rapidly rising paraprotein of >25% or >5g/l over 3 months
  4. splenomegaly
  5. bulky lymphadenopathy
  6. B symptoms or paraneoplastic phenomena, which, in the opinion of the investigator are the result of progressive WM.
* Life expectancy >12 months
* ECOG < 3
* Able to provide informed consent
* Ability to understand the requirements of the study, provide written informed consent, including consent for the use and disclosure of research-related health information, and comply with the protocol procedures, including required study visits.
* Subjects of child bearing potential must agree to use effective contraception throughout the study and for 3 months after the last dose of belimumab

Exclusion Criteria:

* Prior therapy with belimumab.
* Pregnant or breast feeding
* Chemotherapy, immunotherapy or biological therapy within 4 weeks of enrolment. Therapeutic plasma exchange can continue- see section 3.1.4.
* Creatinine clearance (calculated by Cockcroft-Gault) < 60ml/min
* Bilirubin >2x ULN, ALT >2x ULN.
* History of an allergic or anaphylactic reaction to parenteral administration of contrast agents, human or murine proteins or monoclonal antibodies, a history of severe allergic reaction to drugs, food, or insects requiring medical intervention, or a history of hypersensitive triad (having all 3 features of allergic rhinitis with nasal polyps, asthma, and aspirin sensitivity).
* Prior opportunistic infection including tuberculosis or atypical mycobacterial infection, multi-dermatome Herpes Zoster or Pneumocystis pneumonia or invasive fungal infection (not including oral or vaginal candidiasis or superficial dermatophytes) .
* Active infection with hepatitis B, hepatitis C or HIV or historically positive test or test positive at screening for HIV antibody, hepatitis B surface antigen, or hepatitis C antibody.
* History of organ transplant (eg, heart, lung, kidney, liver) or hematopoietic stem cell/marrow transplant.
* Planned surgical procedure during the treatment period of this study or a history of any other medical disease (eg, cardiopulmonary), laboratory abnormality, or condition that, in the opinion of the principal investigator, makes the subject unsuitable for the study.
* Hospitalization for treatment of infection within 60 days of Day 1.
* Use of parenteral (IV or IM) antibiotics (antibacterials, antivirals, anti-fungals, or anti parasitic agents) within 60 days of Day 1.
* Current drug or alcohol abuse or dependence, or a history of drug or alcohol abuse or dependence within 364 days prior to Day 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2009-11; Primary Completion 2012-06 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
Safety of Belimumab infusions in symptomatic WM | Patients are assessed every 28 days while on treatment

SECONDARY OUTCOMES:
Reduction of IgM paraprotein | Serum Immunoglobulins will be tested every 28 days
Reduction of splenomegaly and/or lymphadenopathy | This will be tested every 28 days
Improvement in anaemia | Patients will be assessed every 28 days while on treatment
Correlate the degree of response with Belimumab levels | Pharmacokinetics will be performed on days 1, 15, 56, 168, 364

CONTACTS AND LOCATIONS:
Overall Officials: David Ritchie, Principal Investigator — The Peter MacCallum Cancer Centre; Andrew Spencer, Principal Investigator — The Alfred
Locations (2):
- Australia (2):
  - The Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Alfred Health, Melbourne, Victoria

REFERENCES:
- [Background] Cheema GS, Roschke V, Hilbert DM, Stohl W. Elevated serum B lymphocyte stimulator levels in patients with systemic immune-based rheumatic diseases. Arthritis Rheum. 2001 Jun;44(6):1313-9. doi: 10.1002/1529-0131(200106)44:63.0.CO;2-S. PMID 11407690
- [Background] Elsawa SF, Novak AJ, Grote DM, Ziesmer SC, Witzig TE, Kyle RA, Dillon SR, Harder B, Gross JA, Ansell SM. B-lymphocyte stimulator (BLyS) stimulates immunoglobulin production and malignant B-cell growth in Waldenstrom macroglobulinemia. Blood. 2006 Apr 1;107(7):2882-8. doi: 10.1182/blood-2005-09-3552. Epub 2005 Nov 22. PMID 16304043
- [Background] Furie R, Stohl W, Ginzler EM, Becker M, Mishra N, Chatham W, Merrill JT, Weinstein A, McCune WJ, Zhong J, Cai W, Freimuth W; Belimumab Study Group. Biologic activity and safety of belimumab, a neutralizing anti-B-lymphocyte stimulator (BLyS) monoclonal antibody: a phase I trial in patients with systemic lupus erythematosus. Arthritis Res Ther. 2008;10(5):R109. doi: 10.1186/ar2506. Epub 2008 Sep 11. PMID 18786258
- [Background] Gross JA, Dillon SR, Mudri S, Johnston J, Littau A, Roque R, Rixon M, Schou O, Foley KP, Haugen H, McMillen S, Waggie K, Schreckhise RW, Shoemaker K, Vu T, Moore M, Grossman A, Clegg CH. TACI-Ig neutralizes molecules critical for B cell development and autoimmune disease. impaired B cell maturation in mice lacking BLyS. Immunity. 2001 Aug;15(2):289-302. doi: 10.1016/s1074-7613(01)00183-2. PMID 11520463
- [Background] Gross JA, Johnston J, Mudri S, Enselman R, Dillon SR, Madden K, Xu W, Parrish-Novak J, Foster D, Lofton-Day C, Moore M, Littau A, Grossman A, Haugen H, Foley K, Blumberg H, Harrison K, Kindsvogel W, Clegg CH. TACI and BCMA are receptors for a TNF homologue implicated in B-cell autoimmune disease. Nature. 2000 Apr 27;404(6781):995-9. doi: 10.1038/35010115. PMID 10801128
- [Background] Halpern WG, Lappin P, Zanardi T, Cai W, Corcoran M, Zhong J, Baker KP. Chronic administration of belimumab, a BLyS antagonist, decreases tissue and peripheral blood B-lymphocyte populations in cynomolgus monkeys: pharmacokinetic, pharmacodynamic, and toxicologic effects. Toxicol Sci. 2006 Jun;91(2):586-99. doi: 10.1093/toxsci/kfj148. Epub 2006 Mar 3. PMID 16517838
- [Background] Kimby E, Treon SP, Anagnostopoulos A, Dimopoulos M, Garcia-Sanz R, Gertz MA, Johnson S, LeBlond V, Fermand JP, Maloney DG, Merlini G, Morel P, Morra E, Nichols G, Ocio EM, Owen R, Stone M, Blade J. Update on recommendations for assessing response from the Third International Workshop on Waldenstrom's Macroglobulinemia. Clin Lymphoma Myeloma. 2006 Mar;6(5):380-3. doi: 10.3816/CLM.2006.n.013. PMID 16640813
- [Background] Mackay F, Woodcock SA, Lawton P, Ambrose C, Baetscher M, Schneider P, Tschopp J, Browning JL. Mice transgenic for BAFF develop lymphocytic disorders along with autoimmune manifestations. J Exp Med. 1999 Dec 6;190(11):1697-710. doi: 10.1084/jem.190.11.1697. PMID 10587360
- [Background] Petri M, Stohl W, Chatham W, McCune WJ, Chevrier M, Ryel J, Recta V, Zhong J, Freimuth W. Association of plasma B lymphocyte stimulator levels and disease activity in systemic lupus erythematosus. Arthritis Rheum. 2008 Aug;58(8):2453-9. doi: 10.1002/art.23678. PMID 18668552
- [Background] Rennert P, Schneider P, Cachero TG, Thompson J, Trabach L, Hertig S, Holler N, Qian F, Mullen C, Strauch K, Browning JL, Ambrose C, Tschopp J. A soluble form of B cell maturation antigen, a receptor for the tumor necrosis factor family member APRIL, inhibits tumor cell growth. J Exp Med. 2000 Dec 4;192(11):1677-84. doi: 10.1084/jem.192.11.1677. PMID 11104810
- [Background] Scapini P, Carletto A, Nardelli B, Calzetti F, Roschke V, Merigo F, Tamassia N, Pieropan S, Biasi D, Sbarbati A, Sozzani S, Bambara L, Cassatella MA. Proinflammatory mediators elicit secretion of the intracellular B-lymphocyte stimulator pool (BLyS) that is stored in activated neutrophils: implications for inflammatory diseases. Blood. 2005 Jan 15;105(2):830-7. doi: 10.1182/blood-2004-02-0564. Epub 2004 Sep 9. PMID 15358625
- [Background] Scapini P, Nardelli B, Nadali G, Calzetti F, Pizzolo G, Montecucco C, Cassatella MA. G-CSF-stimulated neutrophils are a prominent source of functional BLyS. J Exp Med. 2003 Feb 3;197(3):297-302. doi: 10.1084/jem.20021343. PMID 12566413
- [Background] Schiemann B, Gommerman JL, Vora K, Cachero TG, Shulga-Morskaya S, Dobles M, Frew E, Scott ML. An essential role for BAFF in the normal development of B cells through a BCMA-independent pathway. Science. 2001 Sep 14;293(5537):2111-4. doi: 10.1126/science.1061964. Epub 2001 Aug 16. PMID 11509691
- [Background] Schneider P, Takatsuka H, Wilson A, Mackay F, Tardivel A, Lens S, Cachero TG, Finke D, Beermann F, Tschopp J. Maturation of marginal zone and follicular B cells requires B cell activating factor of the tumor necrosis factor family and is independent of B cell maturation antigen. J Exp Med. 2001 Dec 3;194(11):1691-7. doi: 10.1084/jem.194.11.1691. PMID 11733583
- [Background] Yan M, Marsters SA, Grewal IS, Wang H, Ashkenazi A, Dixit VM. Identification of a receptor for BLyS demonstrates a crucial role in humoral immunity. Nat Immunol. 2000 Jul;1(1):37-41. doi: 10.1038/76889. PMID 10881172
- [Background] Yu G, Boone T, Delaney J, Hawkins N, Kelley M, Ramakrishnan M, McCabe S, Qiu WR, Kornuc M, Xia XZ, Guo J, Stolina M, Boyle WJ, Sarosi I, Hsu H, Senaldi G, Theill LE. APRIL and TALL-I and receptors BCMA and TACI: system for regulating humoral immunity. Nat Immunol. 2000 Sep;1(3):252-6. doi: 10.1038/79802. PMID 10973284
- [Background] Zhang J, Roschke V, Baker KP, Wang Z, Alarcon GS, Fessler BJ, Bastian H, Kimberly RP, Zhou T. Cutting edge: a role for B lymphocyte stimulator in systemic lupus erythematosus. J Immunol. 2001 Jan 1;166(1):6-10. doi: 10.4049/jimmunol.166.1.6. PMID 11123269
- [Background] Locksley RM, Killeen N, Lenardo MJ. The TNF and TNF receptor superfamilies: integrating mammalian biology. Cell. 2001 Feb 23;104(4):487-501. doi: 10.1016/s0092-8674(01)00237-9. No abstract available. PMID 11239407
- [Background] Mackay F, Schneider P, Rennert P, Browning J. BAFF AND APRIL: a tutorial on B cell survival. Annu Rev Immunol. 2003;21:231-64. doi: 10.1146/annurev.immunol.21.120601.141152. Epub 2001 Dec 19. PMID 12427767
- [Background] Thompson JS, Bixler SA, Qian F, Vora K, Scott ML, Cachero TG, Hession C, Schneider P, Sizing ID, Mullen C, Strauch K, Zafari M, Benjamin CD, Tschopp J, Browning JL, Ambrose C. BAFF-R, a newly identified TNF receptor that specifically interacts with BAFF. Science. 2001 Sep 14;293(5537):2108-11. doi: 10.1126/science.1061965. Epub 2001 Aug 16. PMID 11509692
- [Background] Yan M, Wang H, Chan B, Roose-Girma M, Erickson S, Baker T, Tumas D, Grewal IS, Dixit VM. Activation and accumulation of B cells in TACI-deficient mice. Nat Immunol. 2001 Jul;2(7):638-43. doi: 10.1038/89790. PMID 11429549
- [Result] Moore PA, Belvedere O, Orr A, Pieri K, LaFleur DW, Feng P, Soppet D, Charters M, Gentz R, Parmelee D, Li Y, Galperina O, Giri J, Roschke V, Nardelli B, Carrell J, Sosnovtseva S, Greenfield W, Ruben SM, Olsen HS, Fikes J, Hilbert DM. BLyS: member of the tumor necrosis factor family and B lymphocyte stimulator. Science. 1999 Jul 9;285(5425):260-3. doi: 10.1126/science.285.5425.260. PMID 10398604